CLINICAL TRIAL: NCT07014150
Title: An Exploratory Study on the Neoadjuvant Therapy of iIparomlimab and Tuvonralimab Combined With Lenvatinib for Hepatocellular Carcinoma
Brief Title: Neoadjuvant Therapy of iIparomlimab and Tuvonralimab Combined With Lenvatinib for Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QBA001
Record Dates: First submitted 2025-05-29; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma Resectable
Keywords: iIparomlimab and Tuvonralimab; lenvatinib; neoadjuvant therapy; high-risk recurrence; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination medication group (Experimental): Iparomlimab and Tuvonralimab every 21 days up to 3cycles, 7.5mg/kg; Combined with lenvatinib, QD, 8mg/ day for less than 60kg, 12mg/ day for more than 60kg, up to 9 weeks.
  Interventions: Drug: Lenvatinib; Drug: Iparomlimab and Tuvonralimab

INTERVENTIONS:
Drug: Lenvatinib — daily,8mg/ day for less than 60kg, 12mg/ day for more than 60kg, for 9 weeks
Drug: Iparomlimab and Tuvonralimab — 7.5mg/kg, every 3 weeks, for 3cycles.

SUMMARY:
The goal of this clinical trial is to learn if the neoadjuvant therapy of iIparomlimab and Tuvonralimab plus lenvatinib works to treat hepatocellular carcinoma(HCC) patients with high risk of recurrence. It will also learn about the safety of the combination of iIparomlimab and Tuvonralimab plus lenvatinib. The main questions it aims to answer are:

Does the combination therapy improve the major pathological response rate and reduce the risk of disease recurrence or progression in HCC patients? What medical problems do participants have when taking this combination regimen? Researchers will compare this combination to previous studies to evaluate its efficacy and safety in managing HCC.

Participants will:

Take iIparomlimab and Tuvonralimab every 3 weeks for three times and lenvatinib everyday for 9 weeks.

Visit the clinic once every 3 weeks for checkups and tests Keep a diary of their symptoms and the number of times when taking the combination regimen.

DETAILED DESCRIPTION:
This study is a single-center, single-arm, open-label phase II clinical trial, aiming to evaluate the impact of the neoadjuvant treatment regimen ofIparomlimab and Tuvonralimab plus lenvatinib on postoperative recurrence, survival, and drug safety in patients with hepatocellular carcinoma. Primary objective: Major Pathological response Secondary objectives: Efficacy indicators: Pathological complete response, progression-free survival, overall survival, recurrence-free survival, objective response rate, disease control rate. Safety indicators: Vital signs, laboratory parameters, adverse events (AE), serious adverse events (SAE), drug-related AE and SAE, and specific AE of this type of drug. Exploratory objective: To explore the impact of the combined treatment regimen on the tumor immune microenvironment in tumor tissues and peripheral blood of patients.

The target patients are：Patients with hepatocellular carcinoma (HCC) in CNLC stage Ib to IIIa who have at least one of the following high-risk factors for postoperative recurrence: AFP > 400 ng/ml; a single tumor > 5 cm; more than 3 tumors or any one of them > 3 cm; presence of vascular tumor thrombus or tumor adjacent to major vessels, etc.

Researchers will recruit 30 patients who will receive:

Iparomlimab and Tuvonralimab at 7.5 mg/kg administered intravenously every three weeks (q3w) for three cycles; Lenvatinib orally at 8 mg/day for patients weighing ≤60 kg and 12 mg/day for those >60 kg, taken daily for 9 weeks.

Researchers will evaluate whether the combination therapy improve the major pathological response rate and reduce the risk of disease recurrence or progression in HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated in the study and agreed to sign the written informed consent. They had good compliance and cooperated with the follow-up
* Be at least 18 years old at the time of signing the informed consent form, with no gender restrictions.
* Hepatocellular carcinoma diagnosed by histology or imaging
* At least one measurable lesion (according to the requirements of RECIST version 1.1, the long diameter of the measurable lesion on spiral CT scan is ≥10mm or the short diameter of the enlarged lymph node is ≥15mm)
* No systematic treatment has been received before
* CNLC：Ib to IIIa
* There is at least one of the following high-risk factors for postoperative recurrence: AFP>400ng/ml; Single tumor >5cm; The number of tumors is greater than 3 or any one of them is greater than 3cm; There are vascular tumor thrombus or tumors adjacent to large blood vessels, etc.
* The ECOG score was 0-1 within one week before enrollment
* Hematology and organ functions are adequate
* Fertile women: Agree to abstain from sex (avoid heterosexual intercourse) or use contraceptive methods with an annual contraceptive failure rate of less than 1% during the treatment period and for at least 6 months after the last administration

Exclusion Criteria:

* Have received any systemic treatment
* ECOG score >1
* Definite extrahepatic metastasis
* Pregnant women (with a positive pregnancy test before taking the medicine) or lactating women
* Those who are known to be allergic or intolerant to recombinant humanized PD-1 monoclonal antibody drugs and their components (or any excipients)
* Previous or existing grade 3 or above digestive tract fistulas or non-digestive tract fistulas (such as skin) as defined by CTCAE 5.0 criteria
* Major surgical operations (except biopsy) have been performed within 4 weeks before the first study of drug treatment or the surgical incision has not fully healed
* Cardiovascular and cerebrovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction and severe/unstable angina pectoris that occurred within 6 months before enrollment
* Insufficiency of liver and kidney functions, such as jaundice, ascites, and/or bilirubin >3×ULN, creatinine ratio >3.5g/24 hours, etc
* Persistent infection of grade >2 (CTCAE 5.0)
* A history of thromboembolism (including stroke and/or transient ischemic attack) within the past 6 months
* Hypertension that has not been well controlled after antihypertensive drug treatment (systolic blood pressure >160mmHg, diastolic blood pressure >100mmHg)
* An active autoimmune disease or a history of autoimmune diseases in the past two years
* Active central nervous system (CNS) metastases and/or cancerous meningitis
* Be ready or have received organ or allogeneic bone marrow transplants before
* Known history of active tuberculosis (Mycobacterium tuberculosis)
* A history of gastrointestinal bleeding within the past 6 months or a clear tendency towards gastrointestinal bleeding
* History of human immunodeficiency virus (HIV) infection
* Positive for active hepatitis B or hepatitis C and has not received regular treatment. During the screening period, HBV DNA≥2000 IU/ml (or ≥104 copy number /ml), entecavir must be used to reduce it to <2000 IU/ml (or < 104 copy number /ml) before enrollment
* There is drug abuse; Or any medical, psychological or social conditions that may affect the research, cause unstable patient compliance, or even endanger patient safety
* Unresolved toxicity of grade > 1 due to any previous treatment/procedure (CTCAE 5.0, excluding alopecia, anemia, and hypothyroidism).
* Patients with objective evidence of severe lung function impairment in the past or at present, such as a history of severe pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, and drug-related pneumonia
* Received treatment with potent CYP3A4 inhibitors within 7 days before participating in the study
* Accompanied by other malignant tumors, but having had other untreated malignant tumors in the past (within 5 years) or simultaneously, for cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the breast and carcinoma in situ of the cervix, treated superficial bladder cancer and prostate adenocarcinoma that has undergone surgical treatment and whose PSA tumor markers are within the normal range.
* After a comprehensive assessment of the patient's condition by the researchers, it was determined that they were not suitable to participate in this research
* Participate in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological response | after surgery immediately

SECONDARY OUTCOMES:
Overall survival | 12 months after the last subject is enrolled
Recurrence free survival | 12 months after the last subject is enrolled
Disease control rate | From enrollment to the end of treatment at 9 weeks
objective remission rate | From enrollment to the end of treatment at 9 weeks
Progression free survival | 12 months after the last subject is enrolled
Pathological complete response | after surgery immediately
Safety evaluation | From enrollment to the end of treatment at 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences，Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
contact with investivator

REFERENCES:
- [Background] Zhao Y, Ma Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Hao Y, Chen J, Zhang G, Qu S, Li Y, Feng W, Yang M, Liu B, Ouyang W, Liang J, Yu Z, Kang X, Xue S, Yang G, Yan W, Yang Y, Liu Z, Peng Y, Fanslow B, Huang X, Zhang L, Zhao H. First-in-human phase I/Ib study of QL1706 (PSB205), a bifunctional PD1/CTLA4 dual blocker, in patients with advanced solid tumors. J Hematol Oncol. 2023 May 8;16(1):50. doi: 10.1186/s13045-023-01445-1. PMID 37158938
- [Background] Lou, H. et al. Efficacy and safety of iparomlimab and tuvonralimab in previously treated patients with recurrent or metastatic cervical cancer: a multicenter, open-label, single-arm, phase 2 clinical trial (DUBHE-C-206). Int. J. Gynecol. Cancer 34, (2024)